CLINICAL TRIAL: NCT06266390
Title: Engaging the Subgenual Cingulate With Brain Stimulation for Depression
Brief Title: Individualized (fMRI-guided) TMS Treatment for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Desmond Oathes, Associate Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 855007; 1R61MH135428 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-02-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Depression; Major Depressive Disorder; Persistent Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; Brain Imaging; Brain Stimulation; Depression; TMS; fMRI; non-invasive brain stimulation; TMS treatment; TMS for depression; individualized treatment
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will receive rTMS to one of two targets. Participants will be randomly assigned to receive the TMS treatment intervention in one of two target conditions: half to their positive sgACC correlation target, while the remaining half to their negative sgACC correlation target.
Who Masked: Participant
Masking Description: Participants will not be informed on which target they have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Positive Correlation Target (Active Comparator): TMS treatment will be administered using a TMS target positively correlated with the sgACC.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Anticorrelation Target (Active Comparator): TMS treatment will be administered using a TMS target anticorrelated with the sgACC.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — The TMS intervention will involve two sets of Intermittent Theta-Burst Stimulation (iTBS) delivered every weekday for 4-6 weeks. Each iTBS set consists of 40 trains and a total of 1200 pulses, delivered approximately 15 minutes apart, resulting in 2400 pulses per session.

SUMMARY:
The purpose of this study is to investigate the responses of the brain region known as the subgenual anterior cingulate cortex (sgACC) during transcranial magnetic stimulation (TMS) in individuals with depression. Specifically, investigators aim to determine whether the sgACC is engaged when TMS is delivered to specific targets and if the engagement of sgACC changes throughout a full TMS treatment intervention. To achieve this goal, the investigators will employ a combination of TMS and Magnetic Resonance Imaging (MRI) procedures.

Study participation will include completing various questionnaires, clinical assessments, receiving a full transcranial magnetic stimulation (TMS) treatment intervention (every weekday for 6 weeks), and undergoing MRI scans, both with and without concurrent TMS.

DETAILED DESCRIPTION:
Interested subjects will be asked to complete multiple questionnaires, a clinical interview, and a TMS demonstration to determine eligibility following the informed consent process.

If determined eligible, participants will proceed to undergo an MRI scan to generate their individualized TMS targets.The subsequent visit will involve the first MRI scanning session with concurrent TMS (TMS/fMRI), referred to as Baseline TMS/fMRI, along with the completion of multiple questionnaires.

Following the Baseline TMS/fMRI session, participants will begin the TMS treatment phase. This phase comprises daily sessions (Monday to Friday) for 6 weeks, during which participants will receive rTMS treatments and complete various surveys.

Midway through and upon completion of the TMS treatment intervention, two additional TMS/fMRI sessions will replicate the procedures conducted during the initial Baseline TMS/fMRI.

Remote follow-up assessments at 1, 6, and 12 months post-treatment will evaluate any enduring improvements in clinical symptoms.

Participants will be compensated for completing study procedures.

ELIGIBILITY:
Inclusion Criteria

1. 18-65 years old
2. DSM-5 diagnosis of major depressive (at least 90%) or persistent depressive disorder (no more than 10%) as per SCID clinical interview.
3. Patient Health Questionnaire-9 (PHQ-9) score = or > than 10
4. Comprehension of instructions in the English language.
5. Capacity to provide informed consent and follow study procedures.
6. Availability for the duration of the study.

Exclusion Criteria

1. Implanted medical devices, metallic implants, or drug infusion pumps that are not MRI-safe (e.g., aneurysm clips, defibrillators, or cochlear implants)
2. History of significant medical events (e.g., stroke, seizures, brain scarring) or neurological/neurodevelopmental conditions (e.g., epilepsy) that are contraindications for TMS and MRI or may adversely affect brain function and data interpretation.
3. Current psychosis, mania, or substance use disorder
4. Prior failed response to full rTMS or ECT/MST trial. Any successful prior treatments are acceptable and support a prognosis that a new rTMS treatment would be worth attempting.
5. Inability to complete an MRI scan (e.g., claustrophobia, inability to remain still for extended periods).
6. Inability to tolerate TMS administration
7. Significant handicaps that would interfere with testing procedures
8. Acute systemic infection, high fever
9. Acute sleep deprivation or medication/substance intoxication or withdrawal (TMS seizure risk)
10. Current use of cyclosporine, tacrolimus, or others that can cause leukoencephalopathy.
11. Pregnancy
12. Dialysis
13. Suicide attempt in past 6 months (safety precaution)
14. Current use of Bupropion (Wellbutrin) above 300 mg, benzodiazepines, lithium, monoamine oxidase inhibitors (MAOIs), and/or high doses of stimulant medication is exclusionary. Note: Exclusionary dosages or medications may be reduced or discontinued under the supervision of a medical provider. Participants must provide documentation confirming that their medical provider has agreed to oversee any medication changes, as abrupt changes can lower the seizure threshold and are contraindicated for TMS.
15. Transportation limits or physical limits to attending daily M-F treatment sessions.
16. Per study physician discretion medications likely to interfere with blood flow or otherwise compromise functional imaging measures.
17. Any other factor that in the investigators' judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from procedure site; unlikely to be able to schedule daily treatment sessions, etc.)

In addition, during this study participants will be asked to:

1. Refrain from substance use (including marijuana and illicit drugs) for the duration of the study
2. Abstain from alcohol for 24 hours before study visits.
3. Maintain a consistent level of caffeine consumption throughout the study period and avoid any significant increases.
4. Not initiate, discontinue, or adjust any psychiatric medications or therapy treatments during the study period.
5. Inform the study team of any new medical treatments or prescribed medications (e.g., antibiotics) to allow for safety review and determination of continued eligibility for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
sgACC Blood Oxygen Level Dependent (BOLD) signal change following single-pulse fMRI-guided TMS (TMS On vs TMS Off) | Single visit (~2 hours)
  This primary endpoint aims to directly assess sgACC engagement during fMRI-guided TMS by comparing sgACC BOLD signal under TMS On and TMS Off conditions. This sgACC BOLD signal change will be defined as sgACC evoked response henceforth.

SECONDARY OUTCOMES:
Change in sgACC evoked response Pre/Post TMS treatment with positive and negative sgACC correlated targets | Up to 7 weeks
  Test the efficacy of positive and negative functionally connected (FC) targets in inducing changes in sgACC evoked response (modulation) before and after TMS treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States